CLINICAL TRIAL: NCT03121157
Title: Multi-component Technology Intervention for African American Emerging Adults With Asthma
Brief Title: Detroit Young Adult Asthma Project
Acronym: DYAAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wayne State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Karen MacDonell, PhD, Principal Investigator, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HL133506-01 (NIH); R01HL133506 (NIH)
Record Dates: First submitted 2017-03-06; First posted 2017-04-20 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Asthma
Keywords: African Americans; Emerging adults; Medication adherence; eHealth
MeSH Terms: conditions — Asthma; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive two sessions of computer-delivered motivational interviewing via CIAS software programmed to target adherence to medications. The intervention group will also receive text messaged adherence reminders between sessions. Both the computer-delivered sessions and text messages will be tailored to the participant using ecological momentary assessment.
  Interventions: Behavioral: Multi-Component Technology Based Intervention
- Control (No Intervention): Control participants complete CIAS-delivered asthma education modules matched for length, location, and method of delivery of the intervention session. Control participants complete each module at their own pace and then complete a short quiz to assess their knowledge. Control participants also receive text messages between intervention sessions. Message content is the same for all control participants and contains general facts about asthma (not tailored). Message timing is not tailored and is sent at the same time every day (4:00 PM--time chosen to avoid AM and PM medication times but to not interfere with sleep and school activities).

INTERVENTIONS:
Behavioral: Multi-Component Technology Based Intervention — The intervention group receives two sessions of computer-delivered MI via software programmed to target adherence to medications and text messaged adherence reminders between sessions. Sessions are provided by an avatar. The intervention engages the youth with the avatar's communication of empathy, optimism, and autonomy support. The intervention focuses the youth on adherence and relevant health behaviors with feedback on adherence, asthma symptoms, and tailored education. Participants are guided in the planning process through goal setting activities. The length of the intervention sessions are about 30 minutes each, with the total duration of the visit (assessment and intervention) lasting about 1.5 hours.
  Other Names: The Detroit Young Adult Asthma Project (DYAAP)
  Arms: Intervention

SUMMARY:
The purpose of the Detroit Young Adult Asthma Project is to test a technology based program to help African American young adults learn to better manage their asthma. Participants will be randomized to a multi-component technology-based intervention (MCTI) targeting asthma medication adherence or to a comparison control condition.

DETAILED DESCRIPTION:
Racial and ethnic minority youth have poorer asthma status than Caucasian youth, even after controlling for socioeconomic variables. Proper use of asthma controller medications is critical in reducing asthma mortality and morbidity. The clinical consequences of poor asthma management include increased illness complications, excessive functional morbidity, and fatal asthma attacks. There are significant limitations in research on interventions to improve asthma management in racial minority populations, particularly minority adolescents and young adults, though illness management tends to deteriorate after adolescence during emerging adulthood, the unique developmental period beyond adolescence but before adulthood. All elements of the proposed study protocol were piloted in an NHLBI-funded pilot study (1R34HL107664-01A1 MacDonell). Results suggested feasibility and acceptability of the study protocol as well as proof of concept. The intervention is now being tested in a larger randomized clinical trial. The proposed study will include 192 African American emerging adults with moderate to severe persistent asthma and low controller medication adherence recruited from clinic and emergency department settings. Half of the sample will be randomized to receive a multi-component technology-based intervention (MCTI) targeting adherence to daily controller medication. The MCTI consists of two components: 1) 2 sessions of computer-delivered motivational interviewing targeting medication adherence, and 2) individualized text messaging focused on medication adherence between the sessions. Text messages will be individualized based on Ecological Momentary Assessment (EMA). The remaining half of participants will complete a series of computer-delivered asthma education modules matched for length, location, and method of delivery of the intervention session. Control participants will also receive text messages between intervention sessions. Message content will be the same for all control participants and contain general facts about asthma (not tailored). Youth will be recruited from the Detroit Medical Center, the only university affiliated medical center in Detroit, Michigan. It is hypothesized that youth randomized to MCTI will show improvements in adherence to medication (primary outcome) and asthma control (secondary outcome) compared to the comparison condition at all post-intervention follow ups (3, 6, 9, and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* African American, moderate to severe persistent asthma requiring daily controller medications, live within 30 miles of study site (Detroit area), be able to complete questionnaires in English, must own or have access to a cell for phone for study duration.

Exclusion Criteria:

* Thought disorder (i.e. schizophrenia, autism), suicidality, or mental retardation, youth with other chronic health conditions or pregnancy requiring ongoing medical intervention (e.g., HIV, Type II Diabetes).

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | Change from baseline at 3, 6, and 12 months
  Daily text messaging, Doser, and self-report

SECONDARY OUTCOMES:
Asthma Control | Change from baseline at 3, 6, and 12 months
  Frequency of asthma symptoms based on self-report
Asthma Control | Change from baseline at 3, 6, and 12 months
  Lung functioning as measured by portable spirometer

CONTACTS AND LOCATIONS:
Locations (1):
- Detroit Medical Center/Wayne State University School of Medicine, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] MacDonell K, Naar S, Gibson-Scipio W, Bruzzese JM, Wang B, Brody A. The Detroit Young Adult Asthma Project: Proposal for a Multicomponent Technology Intervention for African American Emerging Adults With Asthma. JMIR Res Protoc. 2018 May 7;7(5):e98. doi: 10.2196/resprot.8872. PMID 29735474